CLINICAL TRIAL: NCT06260670
Title: Electrographic Flow Mapping Electrogram Validation in Patients With Persistent Atrial Fibrillation (FLOW EVAL-AF)
Brief Title: FLOW EVAL-AF: FLOW Mapping Electrogram VALidation in Patients With Persistent Atrial Fibrillation
Acronym: FLOW EVAL-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablacon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cortex (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP004
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation; Atrial Fibrillation, Persistent; Arrhythmias, Cardiac
Keywords: Electrographic Flow Mapping
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EGF Mapping (Experimental): Subjects will be treated with catheter ablation of atrial fibrillation as is clinically indicated according to standard hospital ablation procedures (pulmonary vein isolation in de novo, pulmonary vein isolation touch-up in redo).
  In addition, subjects will receive electrographic flow mapping (EGF) and concomitant high density mapping to collect electrogram patterns and morphology using both mapping methods.
  Interventions: Device: Electrographic Flow™ Mapping using Ablamap® Software and FIRMap™ Catheter

INTERVENTIONS:
Device: Electrographic Flow™ Mapping using Ablamap® Software and FIRMap™ Catheter — Subjects will receive ElectroGraphic Flow™ (EGF) mapping with Ablamap® Software and a commercially available 64-pole basket mapping catheter (FIRMap™ Catheter, Abbott Laboratories, Abbott park, IL). The FIRMap™ catheter will be inserted into the right and left atrium to acquire 1 minute recordings of electrical signals in several standardized positions, and turn these into electrographic flow (EGF) maps.
  Subjects will receive concomitant high density (HD) electroanatomical mapping of these regions with the commercially available Ensite Precision mapping system and Advisor™ HD Grid mapping catheter (Abbott Laboratories, Abbott Park, IL).
  Other Names: Ablamap® Electrographic Flow Algorithm Technology

SUMMARY:
FLOW EVAL-AF is a prospective, observational, single center pilot trial. The FLOW EVAL-AF trial is designed to identify driver sources in patients with persistent or longstanding persistent AF using EGF mapping and describe the activation patterns observed from concomitant high density mapping of those regions.

DETAILED DESCRIPTION:
It is hypothesized that initiation and propagation of atrial fibrillation (AF) is dependent, at least in part, on rapid atrial stimulation from focal sources. It is debated whether the mechanism of arrhythmogenesis at these foci is abnormal automaticity, triggered activity, microreentry or rotational reentry. However, after activation emerges from these "driver" sites, fibrillatory conduction ensues resulting in the disorganized conduction pattern of AF. Conventional mapping systems can either achieve high spatial resolution by sequential tachycardia beats following a fixed intra-atrial activation pattern (as in macro reentrant atrial flutter), or high temporal resolution with very low spatial resolution achieved through multielectrode basket catheters. Activation mapping in AF with commercially available mapping systems has been unsuccessful in identifying driver sites because atrial activation patterns change on a beat-to-beat basis precluding the use of sequential mapping approaches, and real-time mapping with basket electrodes lacks sufficient resolution to delineate the complex patterns of conduction.

Electrographic Flow (EGF) mapping (AblaMap®, Ablacon, Inc, Wheat Ridge, CO) is a unique method to assess dominant patterns of intra-atrial conduction during ongoing atrial fibrillation and has been previously described. Recordings from a multielectrode basket catheter are analyzed for electrical activation vectors over sequential 2-second segments during a 60 second acquisition period. Patterns of reproducible vector activation are used to identify driver sources for the atrial fibrillation (AF). Multiple sources are often identified in patients with persistent AF. It is anticipated that substrate modification of these source regions will eliminate the AF drivers and result in a favorable response to catheter ablation as shown in a previously published retrospective analysis.

The FLOW EVAL-AF trial is designed to identify driver sources in patients with persistent or longstanding persistent AF using EGF mapping and describe the activation patterns observed from concomitant high density (HD) mapping of those regions. FLOW EVAL-AF is a prospective, observational, single center pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective catheter ablation of AF
* History of persistent or longstanding persistent AF
* Able to provide written informed consent prior to the procedure
* Age ≥18 years

Exclusion Criteria:

* Presence of a permanent pacemaker or other transvenous pacing/defibrillation leads
* Presence of a prosthetic mitral heart valve
* Known reversible causes of AF
* Any cerebral ischemic event (strokes or transient ischemic attacks) which occurred during the 6-month interval preceding the consent date
* History of thromboembolic event within the past 6 months or evidence of intracardiac thrombus at the time of the procedure
* Unable to provide own informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishaki Mehta, MD, Principal Investigator — William Beaumont Hospitals, Royal Oak, MI; Philipp Sommer, MD, Principal Investigator — Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany
Locations (1):
- Herz-und Diabeteszentrum NRW (Clinic of Ruhr University of Bochum), Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kutinsky I, Nilsson KR, Mrlik M, Kong MH, Mehta N, Castellano S. Electrographic flow (EGF) mapping reveals sex-based differences in EGF patterns with women concentrated in phenotypes that benefit from EGF-guided ablation. J Interv Card Electrophysiol. 2026 Jan 7. doi: 10.1007/s10840-025-02184-8. Online ahead of print. PMID 41498861
- [Derived] Sommer P, Castellano S, Ahapov K, Jansen MM, Mehta NK, Kong MH. A single-center trial of electrographic flow mapping and concomitant voltage mapping in sinus rhythm and atrial fibrillation (FLOW EVAL-AF). J Interv Card Electrophysiol. 2024 Nov 27. doi: 10.1007/s10840-024-01946-0. Online ahead of print. PMID 39604766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single Center in Germany
Groups:
- EGF Mapping Group: Subjects with Persistent Atrial Fibrillation who received Electrographic Flow mapping in the context of the FLOW EVAL-AF study.
Period: Overall Study
Arm/Group | EGF Mapping Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EGF Mapping Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 10
Left Atrium Diameter [Mean (Standard Deviation); unit: cm] | 4.6 (0.5)
CHA2DS2-VASc score [Mean (Standard Deviation); unit: units on a scale [scale range: 0-9]] — Tool to describe risk of ischemic stroke in patients with AF. To help guide the decision to treat patients with anticoagulants. Calculated by adding the number of risk factors: Congestive Heart Failure, Hypertension, Age≥75, Diabetes, Stroke/TIA, Vascular Disease, Age 65-74 years and Female Sex. Each risk factor adds a point to the risk score, except for Age ≥ 75 years & Stroke/TIA, which both add 2 points. Score of 0 represents a patient having no additional risk factors. The ESC guidelines considers a score of 1 to be moderate risk and a score ≥ 2 to be high risk. Range: 0 (low) - 9 (high)
  units on a scale [scale range: 0-9] | 2.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Acquisition of EGF Mapping and High Density Mapping
Description: Number of participants with successful acquisition of global electrographic flow (EGF) maps from each of the right and left atria and high density electrogram acquisitions, from at least 3 basket positions in each atrium.
Time Frame: Intraprocedural
Population: Total FLOW EVAL-AF Study Population
Measure: Count of Participants; unit: Participants
Groups:
- EGF Mapping Group: All subjects in the FLOW EVAL-AF study.
Arm/Group | EGF Mapping Group
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Total Number of EGF-Identified Sources
Description: Total number of Active Sources, identified by Electrographic Flow™ (EGF) Mapping, in the total study population.
  EGF mapping uses optical flow algorithms to identify locations in the atrium that produce excitatory waves during ongoing AF, which may be detectable for varying durations of time. Sources with an active prevalence ≥ 25% were quantified as EGF-identified sources in this study.
Time Frame: Intraprocedural
Population: Total FLOW EVAL-AF Study Population
Measure: Number; unit: EGF-identified Sources
Arm/Group | EGF Mapping Group
Number analyzed (Participants) | 10
EGF-identified Sources | 11

ADVERSE EVENTS:
Time Frame: Subject discharge
Description: Adverse Events were collected until subject discharge, up to 1 week.
Arm/Group | EGF Mapping Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT06260670/Prot_SAP_001.pdf